CLINICAL TRIAL: NCT06193304
Title: An Open-label Study to Assess the Absorption Through the Mouth After Three Repeated 50 mg Doses of Eliglustat Solution, Separated by 2-hour Intervals, Held in the Mouth for 30 Seconds With Swishing But Without Ingestion, in Healthy Subjects
Brief Title: A Study to Evaluate Pharmacokinetic Parameters and Safety of Eliglustat Absorption Through the Mouth
Acronym: Acronym
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: PKM14187; U1111-1294-8055 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Gaucher's Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eliglustat (Experimental): Three repeated doses of eliglustat solution, separated by 2-hour intervals, held in the mouth for 30 seconds with swishing but without ingestion
  Interventions: Drug: Eliglustat

INTERVENTIONS:
Drug: Eliglustat — Pharmaceutical form:solution -Route of administration: Oral wihtout ingestion
  Other Names: GZ385660; CERDELGA

SUMMARY:
A study to assess the absorption of eliglustat through the mouth in healthy subjects and the safety of any systemic exposure resulting from oral surface absorption of eliglustat in healthy subjects.

DETAILED DESCRIPTION:
Duration of the study for each subject, not including screening, will be 3 days including follow-up.

ELIGIBILITY:
Inclusion Criteria:

Body weight between 50.0 and 100.0 kg, inclusive, for males, and between 40.0 and 90.0 kg, inclusive, for females, body mass index between 18.0 and 30.0 kg/m2, inclusive.

Having given written informed consent prior to undertaking any study-related procedure.

Certified as healthy by a comprehensive clinical assessment (detailed medical history, complete physical examination, laboratory parameters, and ecg).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.

Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2014-08-25 (Actual); Primary Completion 2014-09-21 (Actual); Study Completion 2014-09-21 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter: Cmax | Multiple timepoints on Day 1
  Maximum plasma concentration observed (Cmax)
Plasma pharmacokinetic (PK) parameter tmax | Multiple timepoints on Day 1
  Time to reach Cmax (tmax)
Plasma pharmacokinetic (PK) parameter AUClast | Multiple timepoints on Day 1
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast (AUClast)
Plasma pharmacokinetic (PK) parameter AUC 0-2h | Multiple timepoints on Day 1
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to 2 hours (h) post dose (AUC0-2h)
Plasma pharmacokinetic (PK) parameter AUC 2-4h | Multiple timepoints on Day 1
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time 2 hours post dose to 4 hours post dose (AUC2-4h)
Plasma pharmacokinetic (PK) parameter AUC 4-6h | Multiple timepoints on Day 1
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time 4 hours post dose to 6 hours post dose (AUC4-6h)
Plasma pharmacokinetic (PK) parameter tlast | Multiple timepoints on Day 1

SECONDARY OUTCOMES:
Treatment emergent adverse events during the study | Up to Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Researsh Unit, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org